CLINICAL TRIAL: NCT05574517
Title: A Comparative Study of Tubeless Percutaneous Nephrolithotomy With or Without Reverse Ureteral Catheter Insertion
Brief Title: Tubeless Percutaneous Nephrolithotomy Without Reverse Insertion of a Ureteral Catheter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of South China (Other)
Responsible Party: Principal Investigator, Li Mingyong, MD, Associate professor, The First Affiliated Hospital of University of South China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USCKF201902K01
Record Dates: First submitted 2022-10-01; First posted 2022-10-10 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Urinary Calculi; Percutaneous Nephrolithotomy
Keywords: Ureteral catheter; Without reverse insertion; Percutaneous nephrolithotomy; Tubeless; Urinary calculi
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to an experimental or control group in parallel.
Who Masked: Participant
Masking Description: A single-blind trial in which participants were unaware of the study group and the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group(group 1) (Experimental): Without reverse insertion of a ureteral catheter in tubeless percutaneous nephrolithotomy.
  Interventions: Procedure: Without reverse insertion of a ureteral catheter
- Control group(group 2) (No Intervention): Traditional tubeless percutaneous nephrolithotomy need reverse insert a ureteral catheter.

INTERVENTIONS:
Procedure: Without reverse insertion of a ureteral catheter — Traditional tubeless percutaneous nephrolithotomy usually need retrograde ureteral catheter insertion. Our intervention is that the tubeless percutaneous nephrolithotomy is executed without reverse insertion of a ureteral catheter.
  Arms: Experimental group(group 1)

SUMMARY:
Percutaneous nephrolithotomy(PCNL) is a surgical method for upper urinary calculi. The advent of tubeless PCNL (without indwelling nephrostomy tube) has been proved to be safe and effective in reducing postoperative discomfort, shortening hospitalization time and reducing hospitalization costs. Traditional tubeless PCNL usually involves retrograde insertion of the ureteral catheter, which may cause many ureteral related surgical complications. However, there are few reports on tubeless PCNL without reverse ureteral catheter insertion. The goal of this study is to explore the safety and effectiveness of the tubeless PCNL without reverse ureteral catheter insertion.

DETAILED DESCRIPTION:
This is a key clinical research project of the University of South China (No. USCKF201902K01). The goal of this study is to comparative the safety and clinical efficacy between the tubeless percutaneous nephrolithotomy without reverse insertion of a ureteral catheter and the traditional tubeless percutaneous nephrolithotomy with reverse insertion of a ureteral catheter in the treatment of upper urinary calculi, and to explore the former' applications. It is a prospective, randomized controlled single center study that is conducted for 2 years anticipatively. The clinic physician is responsible for patient recruitment and allocation and the application of computerized random-number generation. For random allocation, participants are given random numbers. Participants with odd numbers are assigned to experimental group, where they undergo tubeless PCNL without reverse insertion of a ureteral catheter. Participants with even numbers are assigned to control group and undergo tubeless PCNL with reverse insertion of a ureteral catheter. The doctors managing the operations accept participants and execute the surgical treatments. All participants sign clinical-trial informed consent and surgical informed consent during the preoperative conversation. Follow-up observation is conducted for 1 month after surgery. After completion of the study, we collect relevant clinical data from the participants. The primary and secondary outcomes are analyzed and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants who met the the applications of PCNL surgery in the 2019 Chinese Guidelines for the Diagnosis and Treatment of Urological Diseases
* Participants who agree to undergo tubeless PCNL
* The participants' maximum diameter of the stone should be less than 3.5cm

Exclusion Criteria:

* Confirmation by computerized tomography (CT) images and blood biochemical indicators of infectious stones or complex staghorn stones
* Obvious surgical contraindications, such as severe heart and lung insufficiency, abnormal coagulatory function
* Previous PCNL or nephrolithotomy, presence of an indwelling ureteral stent or nephrostomy tube before surgery
* Renal trauma or congenital malformation of the urinary system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of inflammatory indicators after surgery | Hour 3 after the surgery
  Pre- vs. post-operative blood leukocyte counts and neutrophil-ratio difference
Changes in renal bleeding after surgery | Hour 3 after the surgery
  Pre- vs. post-operative difference in hemoglobin and hematocrit values
Changes of renal-function after surgery | Hour 3 after the surgery
  Preoperative and postoperative blood creatinine difference
Pain score after surgery | Hour 3 after the surgery
  According to the Visual Analogue Scale(VAS) to evaluate the score. Scores range from 0 to 10, where 0 represents no pain and 10 represents the highest pain.
Incidence of pneumothorax and hydrothorax | Day 2 after the surgery
  The rate of pneumothorax and hydrothorax after surgery
Incidence of ureteral stone street | Day 2 after the surgery
  The rate of ureteral stone street after surgery

SECONDARY OUTCOMES:
Duration of operation | during the procedure
  From the completion of anesthesia to the end of the suture incision.
Duration of hospital stay | immediately after the discharge
  From the date of admission to the date of discharge.
Hospital costs | immediately after the discharge
  The cost from hospitalization to discharge.
Stone-free rates | Day 2 after the surgery
  Preoperative and postoperative stone dimensions are compared by radiological assessment. Postoperative residual calculi < 4 mm in diameter reflect complete removal of calculi (stone-free rate = 100%).

CONTACTS AND LOCATIONS:
Overall Officials: Mingyong Li, MD, Principal Investigator — The First Affiliated Hospital of University of South China
Locations (1):
- The First Affiliated Hospital of University of South China, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication.
Supporting Information: Study Protocol, ICF
Time Frame: Starting 1 year after publication.
Access Criteria: When proper editing or review requirements are met, the study data will be available from the study manager after the study is completed.

DOCUMENTS (1):
  • Study Protocol (2022-10-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT05574517/Prot_001.pdf